CLINICAL TRIAL: NCT03667963
Title: Effect of Genetic Variation in Starch-digesting Enzymes on Digestibility and Glycemic Index of Rice Prepared in Different Ways
Brief Title: Effect of Genetic Variation in Starch-digesting Enzymes on Digestibility and Glycemic Index of Cold and Hot Rice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Glycemic Index Laboratories, Inc (Industry)
Responsible Party: Principal Investigator, Thomas Wolever, Professor, University of Toronto
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: RIS protocol number 33593
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Carbohydrate Intolerance
MeSH Terms: conditions — Glucose-Galactose Malabsorption | interventions — Glucose; Lactulose

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Salivary Amylase Activity (Other): Glucose Glucose plus lactulose Hot Rice Cold Rice
  Interventions: Other: Glucose; Other: Glucose plus lactulose; Other: Hot Rice; Other: Cold Rice
- High Salivary Amylase Activity (Other): Glucose Glucose plus lactulose Hot Rice Cold Rice
  Interventions: Other: Glucose; Other: Glucose plus lactulose; Other: Hot Rice; Other: Cold Rice

INTERVENTIONS:
Other: Glucose — 50g glucose dissolved in 250ml water
Other: Glucose plus lactulose — 50g glucose plus 10g lactulose dissolved in 250ml water
Other: Hot Rice — Freshly cooked polished rice containing 50g available carbohydrate (approximately 2/3 cup cooked rice) and consumed hot.
Other: Cold Rice — Cooked polished rice containing 50g available carbohydrate (approximately 2/3 cup cooked rice) cooled overnight in a refrigerator and consumed cold.

SUMMARY:
This study evaluates the effect of different methods of preparation (cooked and consumed hot vs cooked, cooled overnight and consumed cold) and variation in the activity of salivary amylase on the glycemic index and carbohydrate digestibility in healthy human subjects. The effect of genetic variation in small intestinal starch digesting enzymes on glycemic index and starch digestibility will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females aged 18-75 years and in good health
* Eligible to receive income in Canada
* Have Ontario Health Insurance Plan or equivalent medical coverage.
* Previous donor of saliva using protocol reference number # 31093 or GIL-1670 (in which subject consents to measurement of salivary amylase activity and genetic variation in AMY1, SI and MGAM genes).
* Salivary amylase activity in the lowest tertile (<50 U/ml) or highest tertile (>105 U/ml) of salivary amylase activity of 40 subjects previously measured.

Exclusion Criteria:

* known history of AIDS, hepatitis, diabetes or a heart condition
* Allergy to rice, canola oil or sesame oil.
* use of medications (including, but not limited to, insulin or other antidiabetic drugs, systemic steroids, antipsychotics, protease inhibitors, antivirals, immunosuppressive agents and drugs affecting gut motility or digestion) or with any condition which might, in the opinion of Dr. Wolever, the Medical Director or GI Labs, either: 1) make participation dangerous to the participant himself (or herself) or to others, or 2) affect the results.
* individuals who cannot or will not comply with the experimental procedures or do not follow the instructions of GI Labs staff related to the safe performance of the experimental procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Glycemic Index (GI) | 0-2 hours
  For each subject, the incremental area under the glucose response curve over 2 hours (iAUC) after each rice test meal is expressed as a percentage of the mean iAUC elicited by the 2 glucose test meals.

SECONDARY OUTCOMES:
Carbohydrate malabsorbed | 0-6 hours.
  For each test meal the sum of breath hydrogen concentrations from the lowest value over 0-3 hours to 6 hours (termed "H"). For each subject the amount of hydrogen per gram malabsorbed carbohydrate (H/g) is calculated as (GL-G)/10 where GL is H after the glucose plus lactose meal and G is H after the glucose meal. The amount of carbohydrate malabsorbed after the hot and cold rice meals, respectively, are HR/Hg and CR/Hg, where HR and Cr are H after the hot and cold rice meals.
Glycemic response | 0-2 hours
  The incremental area under the blood glucose response curve
Breath hydrogen response | 0-6 hours
  Sum of breath hydrogen concentrations from the lowest in the first 3 hours to 6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — President, Medical Director
Locations (1):
- Glycemic Index Laboratories, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolever TMS, El-Sohemy A, Ezatagha A, Zurbau A, Jenkins AL. Neither low salivary amylase activity, cooling cooked white rice, nor single nucleotide polymorphisms in starch-digesting enzymes reduce glycemic index or starch digestibility: a randomized, crossover trial in healthy adults. Am J Clin Nutr. 2021 Nov 8;114(5):1633-1645. doi: 10.1093/ajcn/nqab228. PMID 34293081